CLINICAL TRIAL: NCT00625105
Title: Using Heart Rate Variability Biofeedback to Improve Attention and Memory in PTSD+ Combat Veterans
Acronym: HRVB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: William Jennings Bryan Dorn VA Medical Center (U.S. Federal Agency)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, J.P. Ginsberg, Ph.D., Principal Investigator, William Jennings Bryan Dorn VA Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: JPG001
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biofeedback (Active Comparator): HRV coherence biofeedback procedure
  Interventions: Behavioral: Biofeedback
- Sham intervention (Sham Comparator): Passive monitor viewing
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Biofeedback

SUMMARY:
This study will test the effectiveness of Heart Rate Variability (HRV) Biofeedback as a therapeutic tool in the reduction of everyday memory problems routinely experienced by combat veterans with Posttraumatic Stress Disorder (PTSD). The study is innovative in three ways: (1) through its investigation of the clinical use of a novel PTSD treatment technology, (2) by focusing on the understudied aspect of the daily functioning of PTSD veterans, and, (3) by investigating a heretofore untested application of biofeedback for PTSD induced deficits in attention (ATTN) and immediate memory (IM). Though HRV Biofeedback has proven successful for several applications in the general population, the idea that deficits in ATTN/IM in combat veterans with PTSD can be remedied by normalization of HRV has not yet been tested empirically. HRV is functionally incorporated into attentional processes, essentially operating as an index of autonomic flexibility and the ability to self-regulate in response to stimulation from the environment. Low HRV occurs in patients with PTSD, General Anxiety Disorder, and Coronary Artery Disease, and is correlated with negative affect and hostility. HRV Biofeedback training has been shown to be effective in increasing HRV in these groups of patients, as well as improving psychological well-being and physiological function in patients with Depression, Fibromyalgia, and Cardiovascular Disease. Therefore, the interrelationship between HRV and ATTN/IM problems in PTSD+ Combat veterans warrants further investigation. If HRV Biofeedback significantly improves ATTN/IM in these subjects, then it can be offered to VA clinicians treating combat PTSD as an effective new treatment tool.

ELIGIBILITY:
Inclusion Criteria:

* OIF/OEF veterans with PTSD

Exclusion Criteria:

* Neurologic disorder
* Active substance abuse

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | completion
Attention and immediate memory | completion

CONTACTS AND LOCATIONS:
Locations (1):
- Dorn VA Medical Center, Columbia, South Carolina, United States